CLINICAL TRIAL: NCT03776188
Title: Prospective Registry for Trans-Orifice Endoscopic Suturing Applications
Brief Title: Endoscopic Suturing (ES) Registry
Status: Completed | Type: Observational
Sponsor: American Gastroenterological Association (Other)
Collaborators: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ES Registry 2-682-101
Record Dates: First submitted 2018-11-03; First posted 2018-12-14 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Surgery
Keywords: Endoscopic Suturing; Bariatric Revision; Stent Fixation; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- no groups - observational study: no groups - observational study

SUMMARY:
To determine patient outcomes (survival, additional endoscopic or surgical procedures) with an endoscopic suturing technique at predetermined intervals compared to historical controls when applicable.

To evaluate the efficacy, safety, and durability of trans-orifice endoscopic suturing therapy for revision of bariatric procedures as well as study the safety, efficacy, and durability of preventative fixation of GI endoprosthetics.

DETAILED DESCRIPTION:
To determine patient outcomes (survival, morbidity including hospitalization, additional re-interventions with radiologic, endoscopic or surgical procedures) with endoscopic suturing at predetermined intervals from the last endoscopic suturing procedure or at failure of the endoscopic suturing with conversion to another intervention such as surgery and compared to historical controls when applicable.

To evaluate the efficacy and safety of endoscopic suturing therapy in preventative fixation of stents and bariatric revision.

To collect data on the common use endoscopic suturing therapy in other indications.

This prospective clinical study is a real-world registry and not a randomized controlled trial. Given the conditions commonly treated with endoscopic suturing and the potential lack of equivalent expertise in open, laparoscopic, and trans-oral surgical procedures at all centers, randomization of participants is not possible nor ethical. In addition, there are clinical scenarios where endoscopic therapy with surgical sutures, tissue sealants, and/or endoprosthetics may be appropriate and open and laparoscopic surgical approaches inappropriate from an ethical viewpoint. Given the multitude of currently available minimally invasive approaches to repair, it would be unethical to expose and randomize patients who are suitable for more minimally invasive approaches to a more invasive and inherently more morbid approach.

This outcomes study is external to the subject receiving the medical device treatment. Subjects will receive the medical device treatment regardless of study participation and the surgery is not part of this research. Subjects will be consented prior to their procedure, to obtain basic follow-up information. If the subject provides informed consent to participate in the registry, then site staff will follow the participant's clinical data for the period of the registry. Site staff may also contact the subject(s) during their standard clinic visit or via the telephone and obtain information on: overall health, specific events related to any subsequent surgical, endoscopic, or radiologic interventions, and hospitalizations.

The clinical data will be collected during usual procedure follow-ups. This will include recording patient demographics, medications, testing results, comorbidities, body mass index, and reason for clinical care visit. If during the follow-up period, the subject undergoes additional clinically indicated procedures or hospitalizations for procedure related indications then the site will submit this information to the registry.

All procedures and device use will be performed as clinically indicated and as directed by the treating physician. All information requested as part of this registry will be obtained from clinical data obtained as part of study.

ELIGIBILITY:
Inclusion Criteria:

1. Selected to undergo trans-orifice suturing prior to study enrollment
2. Age 18+ years
3. Patient ASA classification I, II, III, including emergency cases
4. Patient willing to provide informed consent, cooperate with post-operative recommendations and follow-up assessment

Exclusion Criteria:

1. Patients who do not meet the clinical criteria for trans-orifice suturing
2. Under age 18 years
3. ASA classification IV
4. Unable to provide informed consent
5. Unable to participate in follow-up assessments
6. Uncorrectable coagulopathy at the time of endoscopic suturing
7. Any terminal disease that limits patient's survival to less than one year

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with a condition that can be treated with trans-orifice endoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Dislocation of Stent - distance | Change at 2 weeks, 30 days, 3 months
  Change in the position measured using distance (centimeters).
Dislocation of Stent - location | Change at 2 weeks, 30 days, 3 months
  Change in the position measured using location. Location options: Bridging the GJ anastomosis, Confined to gastric lumen, Bridging the pylorus, Bridging Lower Esophageal Sphincter
Migration Rate of Stent - placement | Change at 2 weeks, 30 days, 3 months
  Distal from placement over time (yes or no)
Migration Rate of Stent - replaced | Change at 2 weeks, 30 days, 3 months
  Stent replaced or re-structured over time (yes or no)
Migration Rate of Stent - sutures | Change at 2 weeks, 30 days, 3 months
  Number of intact Sutures
Migration Rate of Stent - removal | Change at 2 weeks, 30 days, 3 months
  Days to removal and replacement
Excess Weight Loss | Measured at 2 weeks, 30 days, 3 months, 6 months, 12 months
  Changes in body weight measured in kilograms subsequent to the revisional procedure will be summarized using statistics both in percentage terms using the % excess weight lost and absolute terms.
Total Weight Loss | Measured at 2 weeks, 30 days, 3 months, 6 months, 12 months
  Changes in body weight measured in kilograms subsequent to the revisional procedure will be summarized using statistics both in percentage terms using the % total weight loss and absolute terms.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Maranki, MD, Principal Investigator — Penn State Milton S. Hershey School of Medicine
Locations (11):
- United States (11):
  - University of Arkansas, Little Rock, Arkansas
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Borland Grover Clinic, Jacksonville, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Northwell Health, Manhasset, New York
  - New York Presbyterian Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Methodist Dallas Medical Center, Dallas, Texas